CLINICAL TRIAL: NCT06620770
Title: Impact of the Therapeutic Education Program "living with Chronic Inflammatory Disease Under Biotherapy" on Compliance and Quality of Life of Patients
Brief Title: Impact of the Therapeutic Education Program "living with a Chronic Inflammatory Disease Under Biotherapy" on Patient Compliance and Quality of Life
Acronym: IMPEBIO
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier de Bretagne Sud (Other)
Responsible Party: Sponsor
Other Study IDs: 56LORC_2023_IMPEBIO
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Chronic Inflammatory Disease
Keywords: Biotherapy; Therapeutic education program
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients participating in the therapeutic education program: Patients treated with subcutaneous biotherapy who wish to participate in the therapeutic education program will be included in the intervention group. This program will begin within 3 months of inclusion.
  An initial meeting with a nurse allows for a shared educational assessment. The other days are planned monthly with groups of up to 6 people. A discussion around biotherapies is established by a doctor-nurse pair on theoretical and practical questions. In a second step, questions around nutrition are addressed with the dietician. Mealtime is also a time for discussion with professionals and the group of patients. The third workshop is led by a physical activity teacher. A nurse and a patient partner lead a time dedicated to fatigue management in the form of practical exercises that can be easily reproduced at home.
  Interventions: Other: questionnaires
- Patients who do not wish to participate in the therapeutic education program: Patients treated with subcutaneous biotherapy who do not wish to participate in the therapeutic education program will be included in the control group.
  Patients will be followed by their physicians as usual.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Morisky and SF12 Questionnaires delivery at inclusion, 6, 12 and 18 months

SUMMARY:
Patient therapeutic education programs have been shown to be effective in many specialties, allowing "Improving biological and psychological parameters, allowing patients to improve their health knowledge, therapeutic adherence and sense of personal effectiveness." Several studies have shown that patient knowledge, adherence and satisfaction are better after attending a therapeutic education program.

This multidisciplinary program is presented and offered to all patients with chronic disease treated by subcutaneous biotherapy, followed by dermatologists, rheumatologists and gastroenterologists of the Lorient hospital.

The study aims to demonstrate the benefit of the Patient Therapeutic Education program at GHBS Lorient "living with a chronic inflammatory disease under biotherapy" on treatment adherence, as well as the positive impact on quality of life.

DETAILED DESCRIPTION:
All patients followed up as part of their chronic disease and treated with subcutaneous biotherapy in the dermatology, rheumatology, hepatotherapygastroenterology, will be offered participation in the therapeutic education program by GHBS specialists. Whether they agree to participate or not, doctors will offer them participation in the IMPEBIO study.

Patients treated with subcutaneous biotherapy who do not wish to participate in the program will be included in the control group.

Patients treated with subcutaneous biotherapy who wish to participate in this program will be included in the intervention group. The therapeutic education program will begin within 3 months of inclusion.

If the patient does not object, the Morisky scale and the SF 12 questionnaire will be given to him. It may be assisted with filling if necessary by a clinical researcher.

Patients will first complete the Morisky test, and the quality of life questionnaire SF 12 at inclusion in the IMPEBIO study (J0), then to M6 (6 months), M12 (12 months) and M18 (18 months).

These questionnaires will then be retrieved, anonymized and sent to the investigation department. The analysis of questionnaires will not lead to changes in patient management.

Estimated time to complete the questionnaires is 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* All major patients followed up on GHBS for chronic inflammatory disease treated with S/C biotherapy.
* Patients not opposed to their participation in the research.
* Less than 3 months between inclusion and start of Therapeutic Education Program.

Exclusion Criteria:

* Subcutaneous injection by another person.
* Patients with cognitive impairment.
* Persons of legal age who are the subject of a legal protection (safeguarding of justice, curatorship, guardianship), persons deprived of liberty.
* Pregnant women.
* Persons not covered by social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major patients followed up on GHBS for chronic inflammatory disease treated with S/C biotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Scores of the Morisky scale | 18 months after inclusion
  Comparison of the scores of the Morisky scale in patients with chronic inflammatory disease treated by S/C biotherapy at 18 months after inclusion versus patients who only received nurse consultation.

SECONDARY OUTCOMES:
Scores of the Morisky scale | 6 and 12 months after inclusion
  Comparison of scores on the Morisky scale in patients with chronic inflammatory disease treated by S/C biotherapy at 6 and 12 months after inclusion versus patients who only received nurse consultation.
SF-12 quality of life questionnaire | 6 and 12 and 18 months after inclusion
  Comparison of the SF-12 quality of life questionnaire in patients at 6, 12 and 18 months after inclusion versus patients who only received nurse consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Gall, Principal Investigator — Groupe Hospitalier de Bretagne Sud
Locations (1):
- Groupe Hospitalier de Bretagne Sud, Lorient, France

IPD SHARING:
Plan to Share IPD: Undecided